CLINICAL TRIAL: NCT06742216
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial to Evaluate the Efficacy and Safety of Monosialoganglioside in the Treatment of Acute Ischemic Stroke
Brief Title: Monosialoganglioside in Acute Ischemic Stroke: a Randomized, Blinded and Multicenter Confirmatory Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLGM1-AIS-301
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monosialoganglioside (Experimental): Monosialoganglioside GM1, 200 mg/day, for 12-14 days
  Interventions: Drug: Monosialoganglioside
- Placebo (Placebo Comparator): Placebo, for 12-14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Monosialoganglioside — Monosialoganglioside diluted with 0.9% normal saline 100ml, iv, daily for 12-14 days
  Arms: Monosialoganglioside
Drug: Placebo — Placebo diluted with 0.9% normal saline 100ml, iv, daily for 12-14 days
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, parallel, placebo-controlled trial design is used to evaluate the efficacy and safety of GM1 injection in the treatment of patients with acute ischemic stroke.

It is estimated that 1706 patients will be enrolled and randomly assigned to the treatment group and the placebo control group in a 1:1 ratio. Normally, the duration of this study is approximately 90 days.

Treatment was continued for 12~14 days, and follow-up was conducted until the 90th day from the first dose.

The trial is divided into three phases: screening/baseline phase, treatment phase, and follow-up phase.

Screening/baseline period: After the subjects sign the informed consent form, they enter the screening/baseline period for screening examination.

Treatment period: Qualified subjects are randomly divided into groups in a 1:1 ratio and receive continuous treatment for 12~14 days (12~14 times) with GM1 injection and placebo respectively. During the treatment period, relevant examinations and evaluations required by the protocol will be carried out.

Follow-up period: Subjects who have completed treatment will enter the follow-up period until the 90th day of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old；
* Patients with anterior circulation cerebral infarction; first stroke onset or past stroke without obvious neurological deficit (mRS score≤1)；
* Within 24 hours of onset；
* 7 ≤NIHSS score ≤ 20；
* Signed informed consent.

Exclusion Criteria:

* Patients with hereditary abnormal glucose and lipid metabolism (gangliosidosis, such as Tay-Sachs disease and retinal degeneration);
* Hemorrhagic stroke;
* Disturbance of consciousness (NIHSS1a≥1)，or cerebral arteritis, brain tumor, brain trauma, intracranial infectious diseases;
* Planed endovascular treatment;
* Uncontrolled hypertension: systolic pressure ≥200 mmHg or diastolic pressure ≥110 mmHg;
* Bleeding tendency (except for thrombolysis) or severe bleeding within 3 months;
* Patients with malignant tumor or serious diseases;
* Along with epilepsy, arthritis and other disease, which have effect on neurological assessment;
* History of autoimmune diseases, spinal trauma, various demyelinating diseases, including acute inflammatory demyelinating polyneuropathy (Guillain Barre syndrome);
* Unable or unwilling to cooperate due to mental diseases;
* Abnormal liver and renal function: ALT, AST > 2 times of the upper limit of normal value, or Cr > 1.5 times of the upper limit of normal value；
* Hypersensitivity to monosialoganglioside and excipients of test drug;
* History of drug abuse；
* Pregnant or lactating women, pregnant plan or unwilling to use effective contraception during the trial period;
* Participating in other clinical trials within 3 months;
* Other conditions which are unsuitable for this trial assessed by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1232 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-2 | 90 days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome

SECONDARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-1 | 90 days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Gulou Medical College Affiliated Hospital, Nanjing, China